CLINICAL TRIAL: NCT06604468
Title: A Portable Thoracic Impedance Device for Detecting Pulmonary Congestion in Heart Failure Patients
Acronym: DISPLAID1
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-12000
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
Keywords: bioimpedance; heart failure; diuretic treatment; fluid management
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with congestive heart failure: Patients with a diagnosis of congestive heart failure
  Interventions: Diagnostic Test: Thoracic bioimpedance tomography

INTERVENTIONS:
Diagnostic Test: Thoracic bioimpedance tomography — Data collection using a thoracic bioimpedance tomography device

SUMMARY:
This study investigates a portable thoracic bioimpedance tomography (TBIT) device designed to detect early lung congestion in heart failure patients. The main goal is to evaluate how well the device's measurements match those obtained from lung ultrasound and other imaging techniques. By detecting lung fluid build-up before symptoms worsen, this device could help manage heart failure more effectively outside of hospital settings, potentially improving patient care and reducing hospital admissions. Participants in the study are monitored using this device along with standard imaging methods, and data on heart failure symptoms are collected to understand the device's accuracy and usability.

DETAILED DESCRIPTION:
The primary objective is to determine the correlation between TBIT measurements and B-line scores obtained via portable lung ultrasound, with secondary objectives including correlations with thoracic water content from high-resolution CT scans, heart failure symptoms, and NT-proBNP levels adjusted for renal function. Conducted as a prospective, cross-sectional diagnostic study, the research involves heart failure patients recruited during hospital admissions or outpatient visits at heart failure and nephrology clinics. Data collected include TBIT, ultrasound, and CT imaging results, clinical data on heart failure severity, and symptom questionnaires. The study will assess correlations using statistical models such as Spearman's correlation coefficient and mixed-effects models, aiming to validate TBIT as a non-invasive, cost-effective tool for early detection of pulmonary congestion, potentially improving outpatient management and reducing heart failure-related hospitalizations. Ethical considerations include informed consent, confidentiality measures, and ensuring participant safety, with the study procedures being observational and not altering patient treatment based on TBIT results.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Diagnosed with heart failure, defined by the following criterion: hospitalization or an emergency visit for decompensated heart failure (pulmonary edema) within the last 12 months.

Exclusion Criteria:

* Pregnant women at the time of eligibility evaluation.
* Presence of an implanted electronic device in the thorax, such as a pacemaker or defibrillator.
* Inability to provide informed consent.
* Admission to intensive care or the coronary care unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with congestive heart failure
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Lung congestion | Baseline, week 4, week 8
  Assessed using lung ultrasound over 12 thoracic zones to calculate the B-line score

SECONDARY OUTCOMES:
Thoracic water content | Baseline
  Derived using high resolution CT-scan images
Symptom burden | Baseline, week 4 and week 8
  Assessed using the KCCQ-12 questionnaire
NT-pro-BNP | Baseline, week 4, week 8
  Measurement of NT-pro-BNP

OTHER OUTCOMES:
Episodes of decompensated heart failure | 90 days
  Urgent visit or hospitalisation for worsening of heart failure symptoms requiering diuretic treatment or dialysis

CONTACTS AND LOCATIONS:
Locations (1):
- CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided